CLINICAL TRIAL: NCT07058610
Title: Effect of Amplifi Vein Dilation System Treatment on Radiocephalic AVF Maturation-3
Acronym: Amplifi FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amplifi Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLINP1837
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis
Keywords: Amplifi; Pre-dilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Interventional arm (Experimental): Single arm study
  Interventions: Device: Amplifi Vein Dilation System

INTERVENTIONS:
Device: Amplifi Vein Dilation System — An investigational extracorporeal blood pump and catheter system designed to promote vein dilation prior to AVF creation.

SUMMARY:
This multi-phase clinical study evaluated the safety and performance of the Amplifi Vein Dilation System (Amplifi System) in subjects requiring arteriovenous fistula (AVF) creation. Conducted at a single site outside the United States, subjects were enrolled across multiple phases. The study focused on device-related safety, procedural success, percent change in vein dilation and AVF maturation outcomes.

DETAILED DESCRIPTION:
The Amplifi System was used to promote vein dilation prior to AVF creation. Subjects with ESRD or CKD were treated across three phases of enrollment. The protocol incorporated learnings from earlier phases, including improvements to the device design and procedural protocols. This registration covers all phases of the study (Phase 1-3), with updates planned as new data becomes available.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Indicated for wrist or distal forearm radiocephalic AVF creation based on Investigator's standard practice
* ESRD currently receiving maintenance hemodialysis via a tunneled, cuffed hemodialysis catheter
* Baseline wrist or distal forearm cephalic vein diameter of >= 1.7 mm and < 3.2 mm at the proposed Study AVF creation site, wherein the wrist or forearm cephalic vein at the proposed Study AVF creation site is suitable for Amplifi Distal Outflow Catheter placement and Amplifi System treatment, including:

  * >= 1.7 mm to < 3.2 mm diameter of the wrist or forearm cephalic vein at the proposed Study AVF creation site;
  * patency and continuity of blood flow from the proposed Study AVF creation site centrally to the upper arm at the elbow through at least one or more of: 1) the upper arm cephalic vein; 2) the median cubital vein to the upper arm basilic system; or 3) the perforator vein to the deep venous system; and
  * no occlusion or stenosis > 50% along the course of the forearm cephalic vein and at least one upper arm venous outflow up to the subclavian vein, as determined by duplex ultrasonography
* Estimated forearm hemodialysis needle cannulation zone length > 18 cm after creation of the proposed Study AVF
* At least one patent internal jugular vein suitable for Amplifi Inflow Catheter insertion
* Subject has voluntarily signed written informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to any Amplifi System components (polyurethane, nitinol), iodinated contrast agents, heparin, or apixaban
* Known or suspected active infection at the proposed time of Amplifi System placement
* Known bleeding diathesis, including uncorrected coagulopathy
* Known thrombophilia requiring treatment
* Hemoglobin < 10 g/dL
* Platelet count < 100,000/mm³
* Requirement for continued treatment with antiplatelet agents or anticoagulants other than apixaban during the Amplifi System treatment period
* Known history of patent foramen ovale > 2 mm
* History of recent intracranial or gastrointestinal bleeding
* Documented recent central venous or right atrial thrombus
* History of recent ipsilateral central venous occlusion, > 50% stenosis, angioplasty, or stent placement
* Pregnancy, lactation, or plans to become pregnant during the study
* Unwillingness or inability to comply with protocol-specified procedures or follow-up visits
* Participation in another investigational drug or medical device study that has not completed primary endpoint evaluation, that could clinically interfere with study endpoints, or planned participation in such a study prior to completion of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Rate of AVF Maturation at 2 and 6 Weeks | From post AVF creation to end of 6 weeks follow-up.
Percent Change in Cephalic Vein Diameter and Blood Flow | From baseline, during Amplifi System treatment (minimum daily), and prior to Amplifi System removal and AVF creation]
Mean vein diameter of the cephalic vein and blood flow of brachial artery | 2 and 6 weeks post AVF creation
Percentage of subjects who experience an increase in the cephalic vein diameter of ≥2.7 mm from their baseline measurement, or an increase of >1 mm from baseline, following treatment with the Amplifi System. | From baseline measurement to intra-procedural assessment immediately prior to Amplifi System removal and AVF creation (same procedure day)
Rate of Occurrence of Major Device-Related Adverse Events | from device implantation and up to 30 days from device removal and AVF creation

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT07058610/Prot_000.pdf